CLINICAL TRIAL: NCT05369676
Title: Randomized, Double-blind, Phase Ib Clinical Trial to Evaluate the Safety, Pharmacodynamics, and Pharmacokinetic of SSD8432/ Ritonavir Multiple Doses in Treatment of Adults With Asymptomatic Infection, Mild, and Common Type of COVID-19
Brief Title: To Evaluate SSD8432/ Ritonavir in Adults With COVID-19
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B02B11101-103
Record Dates: First submitted 2022-05-01; First posted 2022-05-11 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: COVID-19 Patients

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SSD8432 dose 1 (Experimental): SSD8432 dose 1/ritonavir or placebo
  Interventions: Drug: SSD8432 dose 1/Ritonavir
- SSD8432 dose 2 (Experimental): SSD8432 dose 2/ritonavir or placebo
  Interventions: Drug: SSD8432 dose 2/Ritonavir

INTERVENTIONS:
Drug: SSD8432 dose 1/Ritonavir — Cohort 1:SSD8432/ritonavir or placebo, on day 1 ~day5，BID；
  Other Names: SIM0417 dose 1/Ritonavir
  Arms: SSD8432 dose 1
Drug: SSD8432 dose 2/Ritonavir — Cohort 2:SSD8432/ritonavir or placebo, on day 1 ~day5，BID；
  Other Names: SIM0417 dose 2/Ritonavir
  Arms: SSD8432 dose 2

SUMMARY:
This is a randomized, double-blind, Phase 1b clinical trial to evaluate the safety, Pharmacodynamics, and Pharmacokinetic of SSD8432 combined with ritonavir tablets in adults with COVID-19.

DETAILED DESCRIPTION:
This is a randomized, double-blinded, placebo-controlled, dose-climbing Phase Ib clinical trial, designed to evaluate the safety, pharmacodynamics, and pharmacokinetics of SSD8432/ ritonavir versus placebo in asymptomatic, mild, and common type adult COVID-19 subjects.

This clinical trial is planned to enroll 32 asymptomatic infected, mild or common type adult COVID-19 subjects, divided into 2 cohorts according to different doses of SSD8432:

Cohort 1: 16 subjects, 12 subjects will receive low-dose SSD8432/ ritonavir, and 4 subjects received placebo; Cohort 2: 16 subjects, 12 subjects will receive high-dose SSD8432/ ritonavir, and 4 subjects received placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤75, male or female.
2. Asymptomatic Infection, Mild, or Common Type of COVID-19.
3. Initial positive test of SARS-Cov-2 within 5 days of randomization.
4. Initial onset of COVID-19 signs/symptoms within 3 days of randomization.
5. The Ct value of SARS-COV-2 nucleic acid test before randomization is ≤ 25, or the Ct value is >25 and sarS-COV-2 serum IgG and IgM are negative.

Exclusion Criteria:

1. Transnasal high-flow oxygen therapy or non-invasive ventilation, invasive mechanical ventilation, or ECMO is required or anticipated to be urgently required.
2. Prior to current disease episode, any confirmed SARS-CoV-2 infection.
3. Known medical history of active liver disease (other than nonalcoholic hepatic steatosis).
4. Receiving dialysis or have known moderate to severe renal impairment.
5. Known human immunodeficiency virus (HIV) infection.
6. Suspected or confirmed concurrent active systemic infection other than COVID-19 that may interfere with the evaluation of response to the study intervention.s.
7. Oxygen saturation of ≤ 93% on room air obtained at rest within 24 hours prior to randomization..
8. Treatment with antivirals against SARS-CoV-2 within 14 days.
9. Current or expected use of any medications or substances that are highly dependent on CYP3A4 for clearance.
10. Concomitant use of any medications or substances that are strong inducers of CYP3A4 are prohibited within 28 days.
11. Has received or is expected to receive COVID-19 monoclonal antibody, convalescent COVID-19 plasma or other prohibited concomitant medication.
12. Females who are pregnant or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2022-08-29 (Actual)

PRIMARY OUTCOMES:
Adverse events | Baseline through Day 28
  Frequency of TEAE

SECONDARY OUTCOMES:
Viral load | Baseline through Day 28
  Changes of viral load compared to the baseline
Time to Sustained Alleviation | Baseline through Day 28
  Time to Sustained Alleviation of Targeted COVID-19 Signs/Symptoms
Proportion of Participants Progressing to a Worsening Status (higher score) | Baseline through Day 28
  WHO clinical progression scale (0 to 10)
Maximum Plasma Concentration [Cmax] | Baseline through Day 5
  Plasma Concentration of SSD8432
Area Under the Plasma concentration-time Curve [AUC] | Baseline through Day 5
  Plasma Concentration of SSD8432

CONTACTS AND LOCATIONS:
Overall Officials: Yumei Yang, Study Director — Jiangsu Xiansheng Pharmaceutical Co., LTD
Locations (1):
- Shenzhen Third People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yao B-F, Yang Y, Xu S-S, Tang B-H, Chen J, Guo Z-J, Hu H-L, Zhang W, Fu S-M, Zhang X-F, Hao G-X, Yang X-M, Song L-L, Ye P-P, Liu L, Zhu S-W, Zheng Y, Zhao W. Model-informed drug development in public health emergency of international concern: accelerating marketing authorization of simnotrelvir. Antimicrob Agents Chemother. 2025 Nov 5;69(11):e0061425. doi: 10.1128/aac.00614-25. Epub 2025 Sep 18. PMID 40965470
- [Derived] Wang F, Xiao W, Tang Y, Cao M, Shu D, Asakawa T, Xu Y, Jiang X, Zhang L, Wang W, Tang J, Huang Y, Yang Y, Yang Y, Tang R, Shen J, Lu H. Efficacy and safety of SIM0417 (SSD8432) plus ritonavir for COVID-19 treatment: a randomised, double-blind, placebo-controlled, phase 1b trial. Lancet Reg Health West Pac. 2023 Jul 11;38:100835. doi: 10.1016/j.lanwpc.2023.100835. eCollection 2023 Sep. PMID 37484496